CLINICAL TRIAL: NCT00759733
Title: Prospective Cohort Evaluation of Cardiac Function With Echocardiography and Serum B-type Natriuretic Peptide (BNP) in Obstetrical Patients With and Without a History of Cardiac Disease
Brief Title: Evaluation Cardiac Function With Echo and BNP in Obstetrical Patients With/Without Cardiac Disease
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Crouse Hospital (Other); Central New York Community Foundation, Inc. (Other)
Responsible Party: Principal Investigator, FolkJ, Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: IRBPHS 5123
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Pregnancy; Heart Diseases
Keywords: pregnancy; heart disease; heart function testing; echocardiography; B-type natriuretic peptide; obstetrical care
MeSH Terms: conditions — Heart Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Pregnant women with a history of cardiac disease (study group)
  Interventions: Procedure: echocardiography; Procedure: blood draw for serum B-type natriuretic peptide
- 2: Pregnant women with no history of heart disease (control group)
  Interventions: Procedure: echocardiography; Procedure: blood draw for serum B-type natriuretic peptide

INTERVENTIONS:
Procedure: echocardiography — A non-invasive assessment of cardiac function using sound waves to create a picture of the pregnant woman's heart. There is no radiation involved.
  Other Names: echocardiogram
Procedure: blood draw for serum B-type natriuretic peptide — A simple, minimally invasive standard blood draw for assessment of serum B-type natriuretic peptide, to be measured in a standard hospital laboratory and recorded for research purposes only
  Other Names: BNP

SUMMARY:
Maternal cardiac disease complicates approximately 2 percent of pregnancies and is the leading cause of non-obstetrical maternal death. Evaluating cardiac function and dysfunction is a complex process requiring skilled clinicians and technology such as ECG, long-term monitoring, and echocardiography. A fast, easily obtained blood test for B-type natriuretic peptide (BNP) has been developed that can give evidence for heart muscle stretch and dysfunction among adults with suspected congestive heart failure. Preliminary experience indicates that ventricular dysfunction among OB patients with a history of heart disease can be detected with this serum assay. A prospective cohort design consisting of two groups of pregnant patients; one with a history of cardiac disease and one without, will be followed over the course of the pregnancies and cardiac function will be measured using echocardiography and serum BNP. It is hoped that the blood test for BNP will be a reliable way to help evaluate OB patients with suspected abnormal heart function.

DETAILED DESCRIPTION:
The incidence of cardiac disease during pregnancy is about 2 percent, and is the leading cause of non-obstetrical maternal mortality (1). Women with known cardiac disease and suspected cardiac dysfunction have been monitored and evaluated during pregnancy, labor, delivery, and post partum with electrocardiogram, long-term rhythm recording, and echocardiogram (2). Physiological changes that occur in normal pregnancy include a 43% increase in cardiac output, 45 to 50% increase in intravascular volume, 14% decrease in serum colloid osmotic pressure, and 28% decrease in the colloid osmotic pressure to pulmonary capillary wedge pressure ratio. These hemodynamic changes are believed to maintain adequate uteroplacental perfusion, meet the increased oxygen and nutritional demands throughout gestation and to protect against sudden hemodynamic changes precipitated by blood loss, decreased venous return to the heart, and hypotension (3).

B-type natriuretic peptide [BNP] is released from ventricular myocardium in response to increased ventricular wall tension or stretch. A rapid assay for the measurement of serum BNP levels has been developed and is in clinical use for the evaluation of dyspnea related to ventricular dysfunction. Serum BNP determination has been described as having a higher level of diagnostic accuracy for congestive heart failure as a cause for dyspnea than any other single historical, physical, or laboratory finding. When used in conjunction with other clinical information, the rapid assay for serum BNP levels is useful in establishing or excluding cardiac dysfunction as a cause for acute onset dyspnea (4). During uncomplicated pregnancy, serum BNP levels remain the same as levels seen in non-pregnant women. Among patients with severe preeclampsia, serum BNP levels have been observed to rise to eight times baseline values. Decreased left ventricular ejection fraction and percentage of fractional shortening within myocardium was observed in the preeclampsia group compared to the normal pregnancy group. The degree of structural and functional change was linearly related to the degree of elevation of cardiac natriuretic peptides, including B-type natriuretic peptide levels (5).

Preliminary clinical experience indicates that serum BNP levels obtained by a commercially available rapid assay method may be related to the degree of ventricular dysfunction among obstetrical patients with acute dyspnea associated with preeclampsia, tocolysis therapy, or an underlying history of cardiopulmonary disease (6). The purpose of this protocol is to determine prospectively if the measurement of serum BNP levels will correlate with cardiac function changes noted on echocardiography and clinically among pregnant women with a history of cardiac disease. This group is to be compared to a group of pregnant women with no history of cardiac disease.

Specific Objectives

The specific objectives of this study include the following:

1. Establish a cohort of subjects that have a history of heart disease that have a diagnosis of cardiac disease, either congenital or acquired, that are pregnant and wish to continue their pregnancies through to delivery.
2. Provide standard obstetrical and cardiac care for these subjects and their fetuses as would be indicated by the type, nature, and degree of cardiac disease present from the first trimester until after delivery.
3. Study interventions to include a series of echocardiograms to begin at the time of pregnancy diagnosis and proceed until the end of the post partum time frame. These studies will take place in the first, second, third trimesters, during labor, two to three days after delivery, and six weeks post partum.
4. With each echocardiogram a serum BNP level will be drawn and measured for correlation with the findings noted on echocardiography.
5. Additional data may be collected if an individual subject were to require additional evaluations with echocardiography and/or BNP serum measurements based on clinical indications.
6. Establish a cohort of control subjects with no history of cardiac disease that will have echocardiography and serum BNP measurements on the same schedule described for subjects with a history of cardiac disease for comparison.
7. At the completion of the study, a description of physiologic changes in cardiac function in the cardiac disease cohort attributable to the subjects' history of cardiac disease versus those attributable to the normal physiologic changes of pregnancy will be available.
8. At the completion of the study, a description of changes in the serum levels of BNP will reflect cardiac dysfunction.

Study Design

This study protocol employs a prospective cohort design. A group of woman with a history of cardiac disease and pregnancy will be identified as potential subjects for a study cohort. Each potential subject will have an initial assessment of her cardiac history, condition, and functional status. A detailed review of her complete medical, surgical, gynecologic, and obstetrical history will be obtained as dictated by standard care. Appropriate management for each potential subject's medical and obstetrical care will be initiated and undertaken by accepted clinical practice. Potential subjects for this cohort will be obstetrical patients either cared for directly by or in consultation with the Regional Perinatal Center, Division of Maternal Fetal Medicine, Department of Obstetrics & Gynecology, SUNY Upstate Medical University.

A second group of women with no history of cardiac disease and pregnancy will also be identified as potential subjects for a control cohort. Each potential subject will also have an initial assessment of her medical, surgical, gynecologic, and obstetrical history as dictated by standard care. Appropriate management for each potential subject's medical and obstetrical care will be initiated and undertaken by accepted clinical practice. Potential subjects for this cohort will be obstetrical patients either cared for directly by or in consultation with the Regional Perinatal Center, Division of Maternal Fetal Medicine, Department of Obstetrics & Gynecology, SUNY Upstate Medical University.

In addition to the management given as part of standard medical and obstetrical care, each subject from both cohorts will have a series of serum BNP measurements and echocardiograms. A serum BNP measurement and echocardiogram will be obtained during the first, second, and third trimesters, during the course of labor or delivery, 48 to 72 hours post-delivery, and 6 to 8 weeks post-delivery. Additional studies will be obtained as indicated by standard clinical indications. Serum BNP measurements will be made through laboratory services available at SUNY Upstate Medical University or Crouse Hospital. Echocardiogram studies will be performed at Cardiology P.C. or Pediatric Cardiology at SUNY Upstate Medical University.

A standard form will be used for each subject to record the results of the serum BNP measurements, results of the maternal echocardiograms, and details of the clinical course experienced by each subject during the course of her pregnancy, labor, delivery, and post-delivery care. Complications related to cardiac function as well as other medical and obstetrical complications will also be recorded. Please see the attached standard data collection form for details.

At the conclusion of the study, a comparison will be made between the cohort of women with cardiac disease and the cohort of woman without cardiac disease. Specific comparison will be made in regard to serum BNP levels, cardiac function as measured on echocardiography, and clinical course.

Statistical Methods, Data Analysis, Interpretation

There are no prior published reports regarding the use of a rapid serum BNP assay to evaluate cardiac function during pregnancy for women with known cardiac disease. From June 1, 2003 to May 31, 2004, the Regional Perinatal Center at SUNY Upstate Medical University provided obstetrical care and consultation for 55 patients with ICD-9 Code 648.63, cardiac disease in pregnancy. Since this is a pilot study, it is anticipated that 20 subjects for the cardiac disease cohort can be followed over the course of 1 to 2 years, along with a control cohort.

Specific measurements that will be obtained by echocardiography and recorded as measures of cardiac function will include:

* Estimated left ventricular ejection fraction
* Estimated left ventricular wall thickness
* Estimated cardiac output
* Right and left atrial chamber volumes
* Right and left ventricular chamber volumes
* Estimated pulmonary artery pressure

Serum BNP measurements will be obtained and recorded as units of picograms/milliliter. Approximately 3-4 milliliters of blood is obtained per assay in a standard lavender-top tube by standard blood sampling methods. The rapid quantitative assay for BNP will be run on the Triage® BNP Test (International) of Biosite Diagnostics, Incorporated, San Diego, California.

Measurements of serum BNP will be correlated with clinical course and objective measures of cardiac function as determined by echocardiography. A linear relationship between the elevation of serum BNP measurement and degree of cardiac dysfunction is expected. Elevated serum BNP and cardiac dysfunction demonstrated on echocardiogram should also correlate with the clinical estimate of NYHA functional status and the degree of congestive failure.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects for the cardiac disease in pregnancy cohort:

1. At least 18 years of age
2. Cardiac disease as per Clark's Maternal Mortality Associated with Pregnancy: Group 1 (mortality less than 1%) atrial septal defect, ventricular septal defect, patent ductus arteriosus, pulmonic or tricuspid valve disease, corrected tetrology of Fallot, bioprosthetic valve, mitral stenosis with NYHA class I and II functional status Group 2 (mortality 5-15%) mitral stenosis with NYHA class III and IV functional status, aortic stenosis, coarctation of aorta without valvular involvement, uncorrected tetrology of Fallot, previous myocardial infarction, Marfan syndrome with normal aorta, mitral stenosis with atrial fibrillation, artificial valve Group 3 (mortality 25-50%) pulmonary hypertension, coarctation of aorta with valvular involvement, Marfan syndrome with aortic involvement (7)
3. Other significant cardiac disease not listed above
4. Other medical disorders, such as diabetes mellitus, chronic hypertension, asthma, other endocrine disorders, et cetera, will be acceptable
5. Diagnosis of a least a single intrauterine pregnancy, multiple gestation acceptable

Potential subjects for pregnancy without cardiac disease cohort:

1. At least 18 years of age
2. Absence of significant cardiac disease, minor cardiac disorders such as mitral valve prolapse without arrythmia
3. Other medical disorders, not directly related to cardiac disease, such as diabetes mellitus, chronic hypertension, asthma, other endocrine disorders et cetera, will be acceptable
4. Diagnosis of at least a single intrauterine pregnancy, multiple gestation acceptable

Exclusion Criteria:

1. Less than 18 years of age
2. Non-viable pregnancy such as a threatened spontaneous miscarriage, or ectopic pregnancy
3. Planned termination of pregnancy, either elective or medically indicated based on history
4. Inability to complete informed consent process or participate in the study protocol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women at least 18 years of age with a history of cardiac disease for the study group and a second group of pregnant women at least 18 years of age with no history of heart disease as controls
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07 (Estimated); Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Assess cardiac function on echocardiography and with serum B-type natriuretic peptide for women with a history of cardiac disease and for a control group with no history of heart disease over the course of pregnancy and compare the groups | first, second, third trimesters of a 40-week pregnancy

SECONDARY OUTCOMES:
Assess for the presence of cardiac dysfunction in the course of a 40-week pregnancy | first, second, third trimesters of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: John J Folk, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (2):
- United States (2):
  - Regional Perinatal Center, Syracuse, New York
  - Cardiology Associates Central New York Physician Office Building, Syracuse, New York

REFERENCES:
- [Background] McAnulty JH, Metcalfe J, Ueland K. Heart disease in pregnancy. Hurst JW, Schlant RC, Rockley CE, et al. (eds) The Heart: Arteries and Veins, 7th Edition. McGraw-Hill Information Services, New York 1990; 1465-1478.
- [Background] Lupton M, Oteng-Ntim E, Ayida G, Steer PJ. Cardiac disease in pregnancy. Curr Opin Obstet Gynecol. 2002 Apr;14(2):137-43. doi: 10.1097/00001703-200204000-00006. PMID 11914690
- [Background] Clark SL, Cotton DB, Lee W, Bishop C, Hill T, Southwick J, Pivarnik J, Spillman T, DeVore GR, Phelan J, et al. Central hemodynamic assessment of normal term pregnancy. Am J Obstet Gynecol. 1989 Dec;161(6 Pt 1):1439-42. doi: 10.1016/0002-9378(89)90900-9. PMID 2603895
- [Background] Maisel AS, Krishnaswamy P, Nowak RM, McCord J, Hollander JE, Duc P, Omland T, Storrow AB, Abraham WT, Wu AH, Clopton P, Steg PG, Westheim A, Knudsen CW, Perez A, Kazanegra R, Herrmann HC, McCullough PA; Breathing Not Properly Multinational Study Investigators. Rapid measurement of B-type natriuretic peptide in the emergency diagnosis of heart failure. N Engl J Med. 2002 Jul 18;347(3):161-7. doi: 10.1056/NEJMoa020233. PMID 12124404
- [Background] Borghi C, Esposti DD, Immordino V, Cassani A, Boschi S, Bovicelli L, Ambrosioni E. Relationship of systemic hemodynamics, left ventricular structure and function, and plasma natriuretic peptide concentrations during pregnancy complicated by preeclampsia. Am J Obstet Gynecol. 2000 Jul;183(1):140-7. doi: 10.1067/mob.2000.105684. PMID 10920322
- [Background] Folk JJ, Lipari CW, Nosovitch JT, Silverman RK, Carlson RJ, Navone AJ. Evaluating ventricular function with B-type natriuretic peptide in obstetric patients. J Reprod Med. 2005 Mar;50(3):147-54. PMID 15841926
- [Background] Clark SL. Structural cardiac disease in pregnancy. Clark SL, Cotton DB, Phelan JP (eds). Critical Care Obstetrics, Medical Economics Books, Oradell, New Jersey 1987; 92-113.